CLINICAL TRIAL: NCT06363292
Title: Phase I Clinical Study to Evaluate the Safety and Tolerability of PRO-231 Ophthalmic Solution Versus VIGAMOXI® on the Ocular Surface of Ophthalmologically and Clinically Healthy Subjects.
Brief Title: Study to Evaluate the Safety and Tolerability of PRO-231 Versus VIGAMOXI® on the Ocular Surface of Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Laboratorios Sophia S.A de C.V. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SOPH231-1221/I
Record Dates: First submitted 2024-04-09; First posted 2024-04-12 (Actual); Results first posted 2025-06-15 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-06

CONDITIONS: Ophthalmological Agent Toxicity; Bacterial Conjunctivitis
MeSH Terms: conditions — Conjunctivitis, Bacterial | interventions — Moxifloxacin

STUDY DESIGN:
Intervention Model Description: Phase I, controlled, comparative, parallel-group, single-blind, single-center, controlled clinical trial.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Single-blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PRO-231 (Experimental): * PRO-231: Moxifloxacin 0.5% Ophthalmic solution.
  * Dosage: 1 drop every 6 hours (3 daily applications [TID], in the right eye).
  * Route of administration: Topical ophthalmic.
  Interventions: Drug: PRO-231
- VIGAMOXI® (Active Comparator): * VIGAMOXI® :Moxifloxacin 0.5% Ophthalmic Solution.
  * Dosage: 1 drop every 6 hours (3 daily applications [TID], in the right eye).
  * Route of administration: Topical ophthalmic.
  Interventions: Drug: VIGAMOXI®

INTERVENTIONS:
Drug: PRO-231 — Moxifloxacin 0.5% Ophthalmic solution.
  Other Names: Moxifloxacin
  Arms: PRO-231
Drug: VIGAMOXI® — Moxifloxacin 0.5% Ophthalmic solution.
  Other Names: Moxifloxacin
  Arms: VIGAMOXI®

SUMMARY:
This is a phase I clinical study evaluating the safety and tolerability of PRO-231 ophthalmic solution through the incidence of unexpected adverse events, incidence of conjunctival hyperemia and chemosis, changes in Best Corrected Visual Acuity (BCVA), changes in ocular surface integrity, compared to VIGAMOXI®.

DETAILED DESCRIPTION:
This is a Phase I, controlled, comparative, parallel-group, single-blind, single-center, controlled clinical trial. The variables to be evaluated include:

Primary (safety):

* Incidence of unexpected adverse events related to the interventions
* Incidence of conjunctival hyperemia and chemosis
* Changes in Best Corrected Visual Acuity (BCVA) assessed with Snellen chart
* Changes in ocular surface integrity using fluorescein staining, using the standard Oxford scale.

Primary (tolerability):

- Changes in the ocular comfort index (OCI) score

Secondary (safety):

- Incidence of unexpected adverse events related to the interventions(excluding conjunctival hyperemia and/or chemosis).

Secondary (tolerability):

- Presence of other ocular symptoms (burning, foreign body sensation, pruritus and lacrimation).

ELIGIBILITY:
Inclusion Criteria:

* Having the ability to voluntarily give their signed informed consent.
* Ophthalmologically and clinically healthy subjects.
* Being able to and willing to comply with scheduled visits, treatment plan, and other study procedures.
* Age between 18 to 45 years.
* Male or female gender.
* Women of childbearing potential who have not undergone Bilateral Tubal Occlusion (BTO [Tubal Ligation]), hysterectomy, or bilateral oophorectomy must ensure continuation (initiated ≥ 30 days prior to signing the informed consent form [ICF]) of the use of a hormonal contraceptive method or intrauterine device (IUD) during the study period.
* Best corrected visual acuity (BCVA) of 20/30 or better in both eyes.
* Corneal staining ≤ grade I on the Oxford Scale.
* Having an intraocular pressure ≥ 10 and ≤ 21 mmHg.

Exclusion Criteria:

* History of hypersensitivity to fluoroquinolones, steroid anti-inflammatories, or any of the components of the drugs under investigation.
* Use of ophthalmic medications from any pharmacological group.
* Use of medications by any other route of administration.
* Use of non-steroidal anti-inflammatory drugs, steroid anti-inflammatory drugs, or antibiotics by any route of administration in the last 30 days.
* History of eye surgery in the last 6 months.
* Use of contact lenses for a period less than two weeks prior to the start of the study, and during the intervention period of this study.
* In the case of women: being pregnant, breastfeeding, or planning to become pregnant within the study period.
* Having participated in any clinical research study 30 days prior to inclusion in this study.
* Having previously participated in this same study.
* History of any chronic-degenerative disease, including Diabetes Mellitus or Systemic Arterial Hypertension.
* Diagnosis of glaucoma or ocular hypertension.
* Known diagnosis of liver or heart disease.
* Presenting active inflammatory or infectious disease at the time of entry into the study.
* Presenting unresolved lesions or traumas at the time of entry into the study.
* Having been subjected to non-ophthalmological surgical procedures in the last 3 months.
* Being or having an immediate family member (e.g., spouse, parent/legal guardian, sibling, or child) who is an employee of the research site or the sponsor, and who directly participates in this study.
* Active smoking (specified as the consumption of cigarettes regardless of the amount and frequency, 4 weeks prior to study inclusion and during the intervention period of this study).
* Active alcoholism (specified as the consumption of alcoholic beverages, regardless of the amount and frequency, 72 hours prior to study inclusion and during the intervention period of this study).

Elimination Criteria

* Withdrawal of their consent to participate in the study (informed consent form).
* Occurrence of a serious adverse event, whether related or not to the interventions, that in the opinion of the principal investigator (PI) and/or the sponsor, could affect the patient's fitness to safely continue with the study procedures.
* Non-tolerability or hypersensitivity to any of the compounds used during the tests -(fluorescein, tetracaine).
* Non-tolerability or hypersensitivity to any of the drugs under investigation.
* Adherence < 80% determined by the subject's diary and corroborated by the final weight of the research products (RP) compared to the initial weight.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 37 (Actual)
Dates: Start 2024-01-30 (Actual); Primary Completion 2024-05-28 (Actual); Study Completion 2024-05-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alejandra Sanchez-Rios, MD, Study Director — Regional Medical Affairs Manager
Locations (1):
- IIMET Investigación e Innovación en Medicina Traslacional, Guadalajara, Jalisco, Mexico

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- PRO-231: * PRO-231: Moxifloxacin 0.5% Ophthalmic solution.
  * Dosage: 1 drop every 6 hours (3 daily applications [TID], in the right eye).
  * Route of administration: Topical ophthalmic.
  PRO-231: Moxifloxacin 0.5% Ophthalmic solution.
- VIGAMOXI®: * VIGAMOXI® :Moxifloxacin 0.5% Ophthalmic Solution.
  * Dosage: 1 drop every 6 hours (3 daily applications [TID], in the right eye).
  * Route of administration: Topical ophthalmic.
  VIGAMOXI®: Moxifloxacin 0.5% Ophthalmic solution.
Period: Overall Study
Arm/Group | PRO-231 | VIGAMOXI®
Started | 18 | 19
Completed | 18 | 19
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | PRO-231 | VIGAMOXI® | Total
Number analyzed (Participants) | 18 | 19 | 37
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 18 | 19 | 37
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 23.55 (4.89) | 25.79 (6.21) | 24.76 (5.69)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 11 | 17
  Male | 12 | 8 | 20
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic | 18 | 19 | 37
Region of Enrollment [Count of Participants; unit: Participants]
  Mexico | 18 | 19 | 37

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Unexpected Adverse Events Related to the Interventions
Description: Any unfavorable medical condition affecting the subject after the administration of the investigation product, related to such intervention. Adverse events where inquired and evaluated in every time point specified in the time frame, however, the final number of adverse events reported throught the entire study was evaluated for each group.
Time Frame: Days 0 (Basal Visit), 3 (Visit 1), 8 (Final Visit) and 12 (Safety Call)
Measure: Number; unit: number of related adverse events
Arm/Group | PRO-231 | VIGAMOXI®
Number analyzed (Participants) | 18 | 19
number of related adverse events | 1 | 4

2. Primary Outcome: Incidence of Conjunctival Hyperemia
Description: Any signs of conjunctival hyperemia in between interventions.
Time Frame: Days 0 (Basal Visit), 3 (Visit 1), and 8 (Final Visit)
Measure: Number; unit: number of patients
Arm/Group | PRO-231 | VIGAMOXI®
Number analyzed (Participants) | 18 | 19
number of patients
  Day 0 (Basal Visit) | 5 | 4
  Day 3 (Visit 1) | 3 | 4
  Day 8 (Final Visit) | 4 | 3

3. Primary Outcome: Changes in Best Corrected Visual Acuity (BCVA)
Description: The BCVA will be evaluated through Snellen chart.
Time Frame: Days 0 (Basal Visit), Days 3 (Visit 1) and 8 (Final Visit)
Measure: Mean (Standard Deviation); unit: Best Corrected Visual Acuity (LogMar)
Arm/Group | PRO-231 | VIGAMOXI®
Number analyzed (Participants) | 18 | 19
Best Corrected Visual Acuity (LogMar)
  Day 0 (Basal Visit) | -0.03 (0.06) | -0.02 (0.07)
  Day 3 (Visit 1) | -0.02 (0.05) | -0.03 (0.05)
  Day 8 (Final Visit) | -0.04 (0.06) | -0.03 (0.07)

4. Primary Outcome: Number of Patients With Any Changes in Grade Measurement of the Integrity of the Ocular Surface (Fluorescein Staining)
Description: Number of patients with any changes in the integrity of the ocular surface using fluorescein staining and evaluated through the Oxford scale compared to baseline. The standard Oxford scale for fluorescein staining has the following criteria: Grade 0- Equal to or less than panel A; Grade I- Equal to or less than panel B, greater than panel A; Grade II- Equal to or less than panel C, greater than panel B; Grade III- Equal or less than panel D, greater than panel C; Grade IV- Equal or less than panel E, greater than panel D; Grade V- Greater than panel E.
Time Frame: Days 0 (Basal Visit), Days 3 (Visit 1) and 8 (Final Visit)
Measure: Count of Participants; unit: Participants
Arm/Group | PRO-231 | VIGAMOXI®
Number analyzed (Participants) | 18 | 19
Participants
  Days 0 (Basal Visit) | 0 | 0
  Days 3 (Visit 1) | 0 | 1
  Day 8 (Final Visit) | 0 | 0

5. Primary Outcome: Changes in the Ocular Comfort Index (OCI) Score Between Interventions.
Description: The Ocular Comfort Index is a questionnaire designed to measure ocular surface irritation. It assesses symptoms related to comfort in cases of ocular surface disorders. The Ocular Comfort Index is composed of 12 items that assess the frequency and intensity symptoms. Each item is scored on a scale from 0 to 6 (never to always, or absent to severe). The total score becomes a linear continuous interval scale, which ranges from 0 (least symptomatic) to 100 (most symptomatic).
  The questionnaire was administered to each research subject, allowing them to respond calmly without any pressure and/or coercion. The results were collected using the Ocular Comfort Index calculator [1], obtaining a logit score and a 0-100 scale score for each subject.
  [1].- M. E. Johnson, "Measurement of Ocular Surface Irritation on a Linear Interval Scale with the Ocular Comfort Index," Investigative Ophthalmology & Visual Science, vol. 48, nº 10, 2007.
Time Frame: Days 0 (Basal Visit), and 8 (Final Visit)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | PRO-231 | VIGAMOXI®
Number analyzed (Participants) | 18 | 19
score on a scale
  Day 0 (Basal Visit) | 25.91 (8.17) | 28.01 (8.60)
  Day 8 (Final Visit) | 19.78 (11.86) | 27.14 (10.22)

6. Secondary Outcome: Incidence of Unexpected Adverse Events (Excluding Conjunctival Hyperemia and Chemosis)
Description: Any unfavorable medical condition affecting the subject after the administration of the investigation product, related to such intervention, excluding conjunctival hyperemia and chemosis. Unexpected adverse events where inquired and evaluated in every time point specified in the time frame, however, the final number of adverse events reported throught the entire study was evaluated for each group.
Time Frame: Days 3 (Visit 1), 8 (Final Visit) and 12 (Safety Call)
Measure: Number; unit: number of unexpected adverse events
Arm/Group | PRO-231 | VIGAMOXI®
Number analyzed (Participants) | 18 | 19
number of unexpected adverse events | 1 | 4

7. Secondary Outcome: To Assess the Tolerability of PRO-231 Ophthalmic Solution
Description: To assess the tolerability of PRO-231 ophthalmic solution applied to the ocular surface, in healthy volunteers, versus VIGAMOXI®, by means of: Presence of ocular symptoms (burning, foreign body sensation, pruritus and lacrimation) between interventions.
Time Frame: Days 3 (Visit 1), 8 (Final Visit)
Measure: Number; unit: ocular symptom events
Arm/Group | PRO-231 | VIGAMOXI®
Number analyzed (Participants) | 18 | 19
ocular symptom events
  Burning Day 0 (Basal Visit) | 0 | 0
  Burning Day 3 (Visit 1) | 4 | 5
  Burning Day 8 (Final Visit) | 3 | 2
  Foreign Body Sensation Day 0 (Basal Visit) | 0 | 0
  Foreign Body Sensation Day 3 (Visit 1) | 1 | 0
  Foreign Body Sensation Day 8 (Final Visit) | 1 | 0
  Pruritus Day 0 (Basal Visit) | 0 | 0
  Pruritus Day 3 (Visit 1) | 3 | 2
  Pruitus Day 8 (Final Visit) | 2 | 2
  Lacrimation Day 0 (Basal Visit) | 0 | 0
  Lacrimation Day 3 (Visit 1) | 0 | 0
  Lacrimation Day 8 (Final Visit) | 0 | 0

ADVERSE EVENTS:
Time Frame: Day 1 (Start of product application) to Day 12 (safety call)
Arm/Group | PRO-231 | VIGAMOXI®
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/19
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/19
Other Adverse Events (participants affected / at risk) | 3/18 | 9/19
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PRO-231 (N=18) | VIGAMOXI® (N=19)
Patient-reported conjunctival redness (Eye disorders) | 2 (2) | 4 (4)
Headache (Nervous system disorders) | 1 (1) | 2 (2)
Dry eye sensation (Eye disorders) | 0 (0) | 1 (1)
Blurred vision (Eye disorders) | 0 (0) | 1 (1)
Heaviness sensation (eyelids) (Eye disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-07-27): https://cdn.clinicaltrials.gov/large-docs/92/NCT06363292/Prot_SAP_000.pdf